CLINICAL TRIAL: NCT00131027
Title: Randomized Controlled Trial to Test Efficacy of High-Dose Methotrexate Consolidation Therapy for BCR-ABL-Negative Acute Lymphoblastic Leukemia in Adults
Brief Title: High-Dose Methotrexate (MTX) for Adult Acute Lymphoblastic Leukemia (ALL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Adult Leukemia Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JALSG ALL202-O
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoblastic Leukemia, Acute
Keywords: acute lymphoblastic leukemia; newly diagnosed; BCR-ABL-negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Daunorubicin; Vincristine; Prednisolone; Asparaginase; Cytarabine; Etoposide; Dexamethasone; Methotrexate; Mercaptopurine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): HD-MTX
  Interventions: Drug: Cyclophosphamide; Drug: Daunorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: L-asparaginase; Drug: Cytarabine; Drug: Etoposide; Drug: Dexamethasone; Drug: Methotrexate; Drug: Mercaptopurine; Drug: Doxorubicin
- B (Active Comparator): ID-MTX
  Interventions: Drug: Cyclophosphamide; Drug: Daunorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: L-asparaginase; Drug: Cytarabine; Drug: Etoposide; Drug: Dexamethasone; Drug: Mercaptopurine; Drug: Doxorubicin; Drug: Methotrexate

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Daunorubicin
Drug: Vincristine
Drug: Prednisolone
Drug: L-asparaginase
Drug: Cytarabine
Drug: Etoposide
Drug: Dexamethasone
Drug: Methotrexate — 3 g/sqm (high dose)
  Arms: A
Drug: Mercaptopurine
Drug: Doxorubicin
Drug: Methotrexate — 0.5 g/sqm (intermediate dose)
  Arms: B

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of high-dose methotrexate consolidation therapy for adult patients with BCR-ABL-negative ALL.

DETAILED DESCRIPTION:
Although the multi-agent chemotherapies in current use produce complete remission for a majority of patients with acute lymphoblastic leukemia (ALL), the prognosis for adult ALL remains discouraging due to a high incidence of relapse. Optimal post-remission therapy, therefore, has been a matter of vital concern. In some pediatric ALL studies, the use of high-dose methotrexate (MTX) as a consolidation therapy, has been shown to improve outcome, however, there has been no randomized controlled trials to test its clinical efficacy in adult ALL. With this concern, the Japan Adult Leukemia Study Group (JALSG) has planned a prospective randomized controlled trial comparing high-dose MTX and intermediate-dose MTX for ALL patients who are negative for BCR-ABL. Those who are positive for BCR-ABL can participate in a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated BCR-ABL-negative ALL
* Age between 25 and 64 years
* Performance status between 0 and 3 (ECOG criteria)
* Adequate functioning of the liver (serum bilirubin level < 2.0 mg/dL); kidneys (serum creatinine level < 2.0 mg/dL); and heart (left ventricular ejection fraction greater than 50% and no severe abnormalities detected on electrocardiograms and echocardiographs).
* Written informed consent to participate in the trial

Exclusion Criteria:

* Uncontrolled active infection
* Another severe and/or life-threatening disease
* Positive for HIV antibody and/or hepatitis B surface (HBs) antigen tests
* Another primary malignancy which is clinically active and/or requires medical interventions
* Pregnant and/or lactating women
* Past history of renal failure

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2002-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
Toxicity | 2 years
The rate of complete remission | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Fumihiko Hayakawa, MD, Study Director — Nagoya University; Tomoki Naoe, MD, Study Chair — Nagoya University
Locations (1):
- Department of Hematology, Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- See also: The JALSG homepage — http://www.jalsg.jp/